CLINICAL TRIAL: NCT02203786
Title: Comparative Effects of a D2 and Mixed D1-D2 Dopamine Antagonist on Gambling and Amphetamine Reinforcement in Pathological Gamblers and Healthy Controls
Brief Title: D1 and D2 Dopamine Receptors in Gambling and Amphetamine Reinforcement
Acronym: HFDEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Daniela Lobo, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 232-2009
Record Dates: First submitted 2014-07-23; First posted 2014-07-30 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Pathological Gambling
Keywords: amphetamine; d1 and d2 receptors; dopamine antagonists; pathological gambling; priming; reinforcement
MeSH Terms: conditions — Gambling | interventions — Haloperidol; Fluphenazine; Dextroamphetamine; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haloperidol (Active Comparator): Subjects randomized to pre-treatment drug sequence 1 (haloperidol on day 1 of each phase), or drug sequence 2 (haloperidol on day 2 of each phase).
  Dose 1: 3 visually identical capsules, each containing 1 mg haloperidol OR 3 visually identical placebo (lactose) capsules
  Dose 2: when participants reach expected peak blood levels for dose 1, they will receive their second dose. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, visually identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 visually identical capsules each containing 10 mg dexedrine.
  Response measured to 15 min session of a commercial slot machine game.
  Interventions: Drug: Haloperidol; Drug: Dexedrine; Drug: Placebo; Behavioral: Slot Machine
- Fluphenazine (Active Comparator): Subjects randomized to pre-treatment drug sequence 1 (fluphenazine on day 1 of each phase), or drug sequence 2 (fluphenazine on day 2 of each phase).
  Dose 1: 3 visually identical capsules, each containing 1 mg fluphenazine OR 3 visually identical placebo (lactose) capsules
  Dose 2: when participants reach expected peak blood levels for dose 1, they will receive their second dose. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, visually identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 visually identical capsules each containing 10 mg dexedrine.
  Response measured to 15 min session of a commercial slot machine game.
  Interventions: Drug: Fluphenazine; Drug: Dexedrine; Drug: Placebo; Behavioral: Slot Machine

INTERVENTIONS:
Drug: Haloperidol — Dose/maximum dose = 3-mg; route = oral. Participants assigned to the haloperidol antagonist group will receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between individual doses).
  Dose 1: 3 visually identical capsules, each containing 1 mg haloperidol.
  Other Names: Teva-Haloperidol; DIN: 00396818; Haldol
  Arms: Haloperidol
Drug: Fluphenazine — Dose/maximum dose = 3-mg; route = oral. Participants assigned to the fluphenazine antagonist group will receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between individual doses).
  Dose 1: 3 visually identical capsules, each containing 1 mg fluphenazine.
  Other Names: APO-Fluphenazine; DIN: 00405345; Prolixin; Permitil
  Arms: Fluphenazine
Drug: Dexedrine — Dose/maximum dose = 20-mg; route = oral. All participants will receive 2 doses (@ 20 mg) during Phase II - sessions 3, 4, with minimum 1 week between individual doses.
  Dose 2: when participants reach expected peak blood levels for dose 1, they will receive their second dose. On sessions 3 and 4 (Phase II), the dose will consist of 2 visually identical capsules each containing 10 mg D-amphetamine.
  Other Names: Dextro-amphetamine sulphate; DIN: 01924516; D-amphetamine
Drug: Placebo — Dose 1: On alternate sessions (1 and 3 or 2 and 4, depending on counterbalancing) participants will receive 3 visually identical placebo (lactose) capsules.
  Dose 2: when participants reach expected peak blood levels for dose 1, they will receive their second dose. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, visually identical to those administered for dose 1.
  Other Names: lactose capsule
Behavioral: Slot Machine — 15 minute play of a commercial slot machine game in bar-simulated laboratory setting.
  Other Names: reward cue

SUMMARY:
To determine if:

1. pathological gambling is similar to psychostimulant addiction as reflected by parallel roles for D1 and D2 receptors in gambling and stimulant reinforcement.
2. these parallel roles are linked with gambling pathology or if they are evident in both gamblers and controls.

DETAILED DESCRIPTION:
BACKGROUND: No previous research appears to have investigated the role of dopamine (DA) D1 or D2 receptors in psychostimulant reinforcement in pathological gamblers. Effects of haloperidol vs. placebo will reveal the role of D2 and the effects of fluphenazine vs. haloperidol will reveal the role of D1 in this process.

OBJECTIVE: This study will begin to define the neurochemistry of Pathological Gambling by examining the roles of dopamine D1 and D2 receptors in gambling reinforcement and psychostimulant reinforcement, and exploring genetic predictors of response to DA probes in Pathological Gambling subjects (subjects) and healthy controls.

METHODS: A double-blind, placebo controlled, counterbalanced between-within design will be employed. Each participant will attend 4 sessions with a minimum of 1 week between sessions to ensure drug washout. Responses to the slot machine will be assessed in sessions 1 and 2 (Phase I), and responses to amphetamine will be assessed in sessions 3 and 4 (Phase II). A second capsule (dummy) will be administered at expected peak levels for each antagonist on sessions 1 and 2 to standardize the procedure across sessions.

Subjective reinforcement self-report scales will be administered at key intervals throughout the study.

HYPOTHESIS: It is hypothesized that haloperidol (3-mg) will increase priming (Desire to Gamble, Gambling word salience) and pleasurable effects (e.g., Enjoyment/Liking) induced by playing a slot machine in Pathological Gambling subjects (N = 40). If gambling and stimulant reinforcement are mediated by common mechanisms, haloperidol will also increase priming and pleasurable effects of amphetamine (20-mg) in Pathological Gambling subjects.

If D1 mediates effects of haloperidol, the mixed D1-D2 antagonist, fluphenazine (fluphenazine; 3-mg) will decrease or not alter responses to the slot machine and amphetamine in Pathological Gambling subjects. If D2 deficits are linked with gambling pathology, haloperidol will not affect slot machine or amphetamine reinforcement in controls (N= 40).

If D1 deficits are linked with gambling pathology, fluphenazine will increase gambling and amphetamine reinforcement in controls, by mitigating undue D1 activation in subjects with high baseline D1 function. If D1 or D2 genes contribute to gambling or amphetamine reinforcement, genotype will predict responses to the manipulations.

ELIGIBILITY:
Inclusion Criteria:

* PATHOLOGICAL GAMBLERS
* otherwise healthy, non-treatment seeking, non-abstinent
* male or female
* ages 19-65
* DSM-IV PG symptom scale score > 5
* SOGS (South Oaks Gambling Screen) score > 5
* nicotine dependence acceptable
* CONTROLS
* healthy
* male or female
* ages 19-65
* DSM-IV PG symptom scale score = 0
* SOGS score = 0
* nicotine dependence acceptable
* must have played slot machine > 5 times

Exclusion Criteria:

* both Pathological Gamblers and Controls
* Axis I psychopathology aside from nicotine dependence (or PG) based on SCID
* Schizotypal or Borderline Personality Disorder based on psychiatric interview
* Family history of schizophrenia or bipolar disorder
* English comprehension below grade 7 level.
* ADS (Alcohol Dependence Scale) > 13 (more than low dependence)
* BDI (Beck Depression Inventory) short form > 10 (more than low depression)
* DAST (Drug Abuse Screening Test) > 4 (possible drug abuse)
* Consumption of > 20/15 (men/women) standard alcoholic drinks/ week (hazardous drinking)
* Smoking > 20 cigarettes/day to help minimize withdrawal symptoms during test phase
* Any prior use of psychostimulant drugs
* Current use of medication that could interact with any of the study medications
* Women who are pregnant or breastfeeding

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Lobo, MD, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] APA (2000) Diagnostic and Statistical Manual of Mental Disorders. IV-TR ed. American Psychiatric Association: Washington, DC.
- [Background] Enggasser JL, de Wit H. Haloperidol reduces stimulant and reinforcing effects of ethanol in social drinkers. Alcohol Clin Exp Res. 2001 Oct;25(10):1448-56. PMID 11696664
- [Background] Holley FO, Magliozzi JR, Stanski DR, Lombrozo L, Hollister LE. Haloperidol kinetics after oral and intravenous doses. Clin Pharmacol Ther. 1983 Apr;33(4):477-84. doi: 10.1038/clpt.1983.65. PMID 6831826
- [Background] Lesieur HR, Blume SB. The South Oaks Gambling Screen (SOGS): a new instrument for the identification of pathological gamblers. Am J Psychiatry. 1987 Sep;144(9):1184-8. doi: 10.1176/ajp.144.9.1184. PMID 3631315
- [Background] Midha KK, McKay G, Edom R, Korchinski ED, Hawes EM, Hall K. Kinetics of oral fluphenazine disposition in humans by GC-MS. Eur J Clin Pharmacol. 1983;25(5):709-11. doi: 10.1007/BF00542363. PMID 6662169
- [Background] Wachtel SR, Ortengren A, de Wit H. The effects of acute haloperidol or risperidone on subjective responses to methamphetamine in healthy volunteers. Drug Alcohol Depend. 2002 Sep 1;68(1):23-33. doi: 10.1016/s0376-8716(02)00104-7. PMID 12167550
- [Background] Wong YN, Wang L, Hartman L, Simcoe D, Chen Y, Laughton W, Eldon R, Markland C, Grebow P. Comparison of the single-dose pharmacokinetics and tolerability of modafinil and dextroamphetamine administered alone or in combination in healthy male volunteers. J Clin Pharmacol. 1998 Oct;38(10):971-8. doi: 10.1002/j.1552-4604.1998.tb04395.x. PMID 9807980
- [Derived] Zack M, Lobo D, Biback C, Fang T, Smart K, Tatone D, Kalia A, Digiacomo D, Kennedy JL. Priming effects of a slot machine game and amphetamine on probabilistic risk-taking in people with gambling disorder and healthy controls. J Clin Exp Neuropsychol. 2023 Feb;45(1):31-60. doi: 10.1080/13803395.2023.2187041. Epub 2023 Mar 15. PMID 36919514
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted for all groups between January 2010 and May 2015
Pre-assignment Details: Pathological Gamblers and healthy Controls were each randomized to receive Haloperidol or Fluphenazine. In each group, treatment sequence (antagonist first, placebo second; or vice versa) was counterbalanced across participants, to control for order effects only (sequence was not a test factor). Two Haloperidol-Controls dropped out after session 1.
Groups:
- Haloperidol - Pathological Gamblers: Dose 1: 3 mg haloperidol (3 capsules @ 1mg each) OR 3 identical placebo capsules on alternate sessions (1 and 3 or 2 and 4, depending on counterbalancing). Dose 2: administered when peak blood levels for dose 1 are reached. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, visually identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 identical capsules each containing 10 mg dexedrine. Response measured to 15 min session of a commercial slot machine game.
  Haloperidol: Dose/maximum dose 3 mg oral. Participants assigned to the haloperidol antagonist group will receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between doses).
  Dexedrine: Dose/maximum dose 20mg oral. All participants will receive 2 doses (@ 20 mg) during Phase II - sessions 3, 4, with minimum 1 week between doses.
- Fluphenazine - Pathological Gamblers: Dose 1: 3 mg fluphenazine (3 capsules @ 1 mg each) OR 3 visually identical placebo capsules on alternate sessions (1 and 3 or 2 and 4, depending on counterbalancing). Dose 2: administered when participants reach peak blood levels for dose 1. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 identical capsules each containing 10 mg dexedrine.
  Response measured to 15 min session of a commercial slot machine game. Participants assigned to the fluphenazine antagonist group will receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between individual doses).
  All participants will receive 2 doses of Dexedrine (@ 20 mg) during Phase II - sessions 3, 4, with minimum 1 week between individual doses.
- Haloperidol - Controls: Dose 1: 3 mg haloperidol (3 capsules @ 1 mg each) OR 3 identical placebo capsules on alternate sessions (1 and 3 or 2 and 4, depending on counterbalancing). Dose 2: administered when peak blood levels for dose 1 are reached. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, visually identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 identical capsules each containing 10 mg dexedrine. Response measured to 15 min session of a commercial slot machine game.
  Haloperidol: Dose/maximum dose 3 mg oral. Participants assigned to the haloperidol antagonist group receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between doses). Dexedrine: Dose/maximum dose 20 mg oral. All participants will receive 2 doses (@ 20 mg) during Phase II - sessions 3, 4, with minimum 1 week between doses.
- Fluphenazine - Controls: Dose 1: 3 mg fluphenazine (3 capsules @ 1mg each) OR 3 visually identical placebo capsules on alternate sessions (1 and 3 or 2 and 4, depending on counterbalancing). Dose 2: administered when participants reach peak blood levels for dose 1. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 identical capsules each containing 10 mg dexedrine.
  Response measured to 15 min session of a commercial slot machine game. Participants assigned to the fluphenazine antagonist group will receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between individual doses).
  All participants will receive 2 doses of Dexedrine (@ 20 mg) during Phase II - sessions 3, 4, with minimum 1 week between individual doses.
Period: Overall Study
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Started | 15 | 15 | 17 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants were above 18 years of age.
Groups:
- Haloperidol - Pathological Gamblers; Fluphenazine - Pathological Gamblers: A total of 15 pathological gamblers were enrolled in this arm.
- Haloperidol - Controls; Fluphenazine - Controls: A total of 15 control subjects were enrolled in this arm.
- Total: Total of all reporting groups
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Full Range); unit: years] | 35.8 [22 to 53] | 33.5 [19 to 49] | 36.1 [19 to 56] | 39.9 [23 to 62] | 36.3 [19 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 7 | 21
  Male | 10 | 11 | 10 | 8 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 11 | 11 | 44
South Oaks Gambling Screen (SOGS) [Mean (Full Range); unit: units on a scale] — Range of possible scores on the SOGS is 0-20. A score of 5 or more indicates "probable pathological gambling" with respect to DSM criteria.
  units on a scale | 11.1 [6 to 18] | 11.7 [5 to 20] | 0 [0 to 0] | 0 [0 to 0] | 5.7 [0 to 20]
Beck Depression Inventory - past 2 weeks [Mean (Standard Deviation); unit: units on a scale] — Measure of depressive symptoms in the past 2 weeks. The scale contains 13 items scored 0-3 in increasing severity (range of possible scores: 0-39). A score of 10 is considered the cut-off for clinically relevant depressive symptoms.
  units on a scale | 4.3 (3.6) | 5.6 (4.5) | 0.9 (1.2) | 1.3 (2.1) | 3.02 (2.85)
Eysenck Impulsivity Scale [Mean (Standard Deviation); unit: units on a scale] — This 19-item yes/no scale measures trait impulsivity. Scores range from 0-19. The normative mean in the general population is 9. The mean score in large samples of people with pathological gambling is also 9.
  units on a scale | 9.2 (4.4) | 8.5 (4.4) | 2.6 (2.1) | 1.6 (2.5) | 5.47 (3.35)
Alcohol Dependence Scale [Mean (Full Range); unit: units on a scale] — This 25-item scale assesses severity of the Alcohol Dependence syndrome. Total scores range from 0-51. A score of 13 corresponds to the 1st quartile and scores from 0-13 are said to indicate low dependence. A score of 9 or more has been associated with alcohol "abuse."
  units on a scale | 1.1 [0 to 4] | 1.6 [0 to 11] | 0.6 [0 to 3] | 0.3 [0 to 4] | 0.9 [0 to 11]
Timeline Followback [Mean (Full Range); unit: number of alcoholic drinks per week] — number of alcoholic drinks per week
  number of alcoholic drinks per week | 2.3 [0 to 8] | 1.5 [0 to 3] | 1.5 [0 to 6] | 1.8 [0 to 5.5] | 1.7 [0 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Subjective Reinforcement Self-report Scales
Description: Self-reported Confidence to Refrain from Gambling (0 - 10) was assessed at test session baseline, before the slot machine and after the slot machine (Phase 1); and before amphetamine and at peak amphetamine (Phase 2). The maximum score (10) denotes complete confidence to refrain from gambling (i.e., NO urge or compulsion to gamble); the minimum score (0) denotes complete lack of confidence to refrain from gambling (i.e., overwhelming urge to gamble). Scores between 10 and 0 denote intermediate confidence to refrain from gambling with LOWER scores denoting less confidence to refrain from gambling -- i.e., GREATER urge or compulsive motivation to gamble. Scores shown are based on single item visual analogue ratings 0-10 from each participant at the specified time point. The mean (SD) of these single item ratings is presented for each sub-group.
Time Frame: At key points in testing: immediately after the slot machine game, and at expected peak subjective-behavioral effects for amphetamine (90-minutes post-capsule administration).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Haloperidol - Controls; Fluphenazine - Controls: A total of 15 controls were enrolled in this arm.
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale
  Drug - Confidence not to gamble after slot machine | 4.8 (2.3) | 4.8 (2.9) | 9.5 (1.1) | 9.3 (1)
  Placebo - Confidence not to gamble after slot mach | 4.2 (2.5) | 4.8 (3.4) | 9 (1.6) | 8.2 (3.4)
  Drug - Confidence not to gamble at peak amphetamin | 5.2 (2.5) | 6.4 (3.2) | 9.8 (0.5) | 9.8 (0.4)
  Plac -Confidence not to gamble at peak amphetamine | 5.5 (2.3) | 5.7 (3.5) | 9.4 (1.1) | 9.3 (2.6)

2. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: Measure changes from baseline, especially physiologic reactivity to the slot machine and amphetamine.
Time Frame: At key points in testing: immediately after the slot machine game (change from session baseline), and at expected peak subjective-behavioral effects for amphetamine (90-minutes post-capsule administration)(change from session baseline).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Number analyzed (Participants) | 15 | 15 | 15 | 15
mm Hg
  Drug-Change in DBP pre-to-post slot machine | 20.2 (24.5) | 22 (23.6) | 15.1 (18.6) | 23.6 (23.8)
  Placebo-Change in DBP pre-to-post slot machine | 22.5 (24.8) | 21.6 (29.3) | 19.1 (24.8) | 19 (23.4)
  Drug-Change in DBP pre-amphetamine to peak amph | 27.2 (24.4) | 32.1 (25.1) | 28.5 (30) | 32.7 (30)
  Placebo-Change in DBP pre-amphetamine to peak amp | 33.6 (29.8) | 35.2 (28) | 26.6 (24.5) | 36.3 (28.3)

3. Secondary Outcome: Cognitive Task Performance
Description: Response time to words (gambling, alcohol, positive affect, negative affect) as a percentage of neutral categorized words (parts of a building). This provides an index of the relative salience of stimuli from these four categories against a baseline of reaction to words with no clinical relevance or emotional valence. Smaller scores indicate faster relative response time to the test stimuli vs. neutral stimuli (i.e., greater salience)
Time Frame: At key points during testing: immediately after the slot machine, at expected peak subjective-behavioral effects for amphetamine (90-minutes post-capsule administration)
Measure: Mean (Standard Deviation); unit: percentage of neutral categorized words
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Number analyzed (Participants) | 15 | 15 | 15 | 15
percentage of neutral categorized words
  post-slots-GAM words under drug | 91.6 (7.9) | 94.0 (6.0) | 94.8 (6.1) | 91.0 (7.9)
  post-slots-ALC words under drug | 95.5 (8.4) | 98.1 (7.6) | 96.5 (6.6) | 93.1 (8.9)
  post-slots POS words under drug | 91.3 (8.7) | 95.3 (7.6) | 93.7 (8.3) | 88.3 (8.4)
  post-slots NEG words under drug | 89.1 (9.5) | 96.5 (7.3) | 89.6 (7.6) | 87.9 (10.2)
  post-slots GAM words under placebo | 91.6 (8.1) | 95.0 (5.3) | 97.2 (7.2) | 92.1 (5.3)
  post-slots ALC words under placebo | 94.8 (6.1) | 99.0 (7.2) | 97.0 (6.5) | 93.3 (4.7)
  post-slots POS words under placebo | 92.7 (8.1) | 94.9 (5.8) | 93.7 (6.1) | 86.8 (10.3)
  post-slots NEG words under placebo | 93.0 (10.4) | 97.2 (13.4) | 92.3 (4.8) | 84.7 (6.7)
  peak AMPH GAM words under drug | 96.7 (3.4) | 95.8 (4.5) | 98.1 (4.5) | 97.0 (5.9)
  peak AMPH ALC words under drug | 101.2 (3.6) | 99.5 (4.6) | 99.1 (3.9) | 100.3 (5.4)
  peak AMPH POS words under drug | 98.2 (3.3) | 98.7 (4.6) | 97.2 (4.7) | 96.3 (4.7)
  peak AMPH NEG words under drug | 99.5 (5.1) | 99.4 (4.8) | 96.8 (3.6) | 98.7 (5.2)
  peak AMPH GAM words under placebo | 95.0 (4.9) | 97.9 (5.8) | 96.8 (2.9) | 96.9 (5.3)
  peak AMPH ALC words under placebo | 99.9 (6.2) | 99.9 (5.3) | 100.2 (4.7) | 97.5 (6.5)
  peak AMPH POS words under placebo | 98.4 (4.7) | 97.7 (5.5) | 97.8 (4.0) | 95.1 (3.3)
  peak AMPH NEG words under placebo | 99.0 (6.5) | 100.0 (3.4) | 98.1 (5.7) | 96.7 (4.4)

4. Secondary Outcome: Betting Behaviour in Laboratory-based Slot Machine Game
Description: Risk taking was operationally defined as credits wagered per spin (mean computed for total spins)
Time Frame: 1x per test session (total of 4 test sessions) for duration of the study: 4 weeks (1 session/week)
Measure: Mean (Standard Deviation); unit: credits/spin on slot machine
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Number analyzed (Participants) | 15 | 15 | 15 | 15
credits/spin on slot machine
  Mean bet under drug | 12.8 (7.2) | 16.0 (10.4) | 11.6 (7.8) | 14.4 (10.0)
  Mean bet under placebo | 10.4 (9.3) | 16.1 (12.4) | 9.5 (10.8) | 12.2 (9.5)

5. Secondary Outcome: Speed of Play on Slot Machine Game
Description: Number of individual spins in a 15-minute slot machine game. Each spin corresponds to one wager.
Time Frame: 15-minutes
Measure: Mean (Standard Deviation); unit: individual spins/15-minutes
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Number analyzed (Participants) | 15 | 15 | 15 | 15
individual spins/15-minutes
  Spins/15-minutes under Drug | 76.9 (35.4) | 78.5 (34.5) | 66.4 (27.9) | 71.8 (30.5)
  Spins/15-minutes under Placebo | 88.6 (32.9) | 68.4 (47.3) | 72.2 (40.5) | 66.7 (31.6)

6. Secondary Outcome: Winnings on Slot Machine Upon Completion of Game
Description: Credits
Time Frame: 15-minutes
Measure: Mean (Standard Deviation); unit: credits
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Number analyzed (Participants) | 15 | 15 | 15 | 15
credits
  Winnings (Final Credit Tally) under drug | 239 (305.1) | 277.8 (300.2) | 449.1 (669.6) | 544.3 (820)
  Winnings (Final Credit Tally) under Placebo | 562.4 (658) | 140.8 (325.7) | 339.2 (427.4) | 215 (214.8)

ADVERSE EVENTS:
Time Frame: Same day as drug administration
Groups:
- Haloperidol - Pathological Gamblers; Haloperidol - Controls: Drug sequence 1 (haloperidol on day 1 of each phase), or drug sequence 2 (haloperidol on day 2 of each phase).
  Dose 1: 3mg haloperidol (3 capsules @ 1mg each) OR 3 identical placebo capsules on alternate sessions (1 and 3 or 2 and 4, depending on counterbalancing). Dose 2: administered when peak blood levels for dose 1 are reached. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, visually identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 identical capsules each containing 10 mg dexedrine.
  Response measured to 15 min session of a commercial slot machine game. Haloperidol: Dose/maximum dose 3mg oral. Participants assigned to the haloperidol antagonist group will receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between doses).
  Dexedrine: Dose/maximum dose 20mg oral. All participants will receive 2 doses (@ 20 mg) during Phase II - sessions 3, 4, with minimum 1 week between doses.
- Fluphenazine - Pathological Gamblers; Fluphenazine - Controls: Drug sequence 1 (fluphenazine on day 1 of each phase), or drug sequence 2 (fluphenazine on day 2 of each phase).
  Dose 1: 3 mg fluphenazine (3 capsules @ 1mg each) OR 3 visually identical placebo capsules on alternate sessions (1 and 3 or 2 and 4, depending on counterbalancing). Dose 2: administered when participants reach peak blood levels for dose 1. On sessions 1 and 2 (Phase I), this will consist of 2 dummy capsules, identical to those administered for dose 1. On sessions 3 and 4 (Phase II), the dose will consist of 2 identical capsules each containing 10 mg dexedrine.
  Response measured to 15 min session of a commercial slot machine game. Participants assigned to the fluphenazine antagonist group will receive 2 doses (@ 3 mg) on alternate sessions (with minimum of 2 weeks between individual doses).
  All participants will receive 2 doses of Dexedrine (@ 20 mg) during Phase II - sessions 3, 4, with minimum 1 week between individual doses.
Arm/Group | Haloperidol - Pathological Gamblers | Fluphenazine - Pathological Gamblers | Haloperidol - Controls | Fluphenazine - Controls
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 2/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haloperidol - Pathological Gamblers (N=15) | Fluphenazine - Pathological Gamblers (N=15) | Haloperidol - Controls (N=15) | Fluphenazine - Controls (N=15)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Mild restlessness which is an expected side effect of haloperidol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No